CLINICAL TRIAL: NCT02553265
Title: Carbidopa in Familial Dysautonomia: Phase-II Study, Investigational New Drug (IND) 117435, Date: 01/07/13
Brief Title: Carbidopa for the Treatment of Excessive Blood Pressure Variability
Acronym: CarbiFD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-00065; FD-R-004772 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Dysautonomia, Familial; Baroreflex Failure Syndrome
Keywords: Familial dysautonomia (HSAN III); Norepinephrine; Sympathetic nervous system; Autonomic nervous system; Blood pressure variability; Hypertension; Carbidopa/Lodosyn; Afferent baroreflex failure; Clinical trial
MeSH Terms: conditions — Dysautonomia, Familial; Hypertension | interventions — Carbidopa; Oxymetholone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo
- Low-Dose Carbidopa (Experimental)
  Interventions: Drug: Carbidopa Low-Dose
- High-Dose Carbidopa (Active Comparator)
  Interventions: Drug: Carbidopa High-Dose

INTERVENTIONS:
Drug: Carbidopa Low-Dose — 300 mg/day
  Other Names: Lodosyn ®, DL-α-methyl-α-hydrazino-3, 4-dihydroxyphenyl-propionic acid, HMD, MK-486
  Arms: Low-Dose Carbidopa
Other: Placebo — A placebo containing an inert substance, in capsule form that does not contain an active drug ingredient.
  Other Names: Placebo control pill
  Arms: Placebo
Drug: Carbidopa High-Dose — 600 mg/day
  Other Names: Lodosyn ®, DL-α-methyl-α-hydrazino-3, 4-dihydroxyphenyl-propionic acid, HMD, MK-486
  Arms: High-Dose Carbidopa

SUMMARY:
The overall study objectives are to determine whether carbidopa (Lodosyn®) is safe and well tolerated and to assess whether it can inhibit catecholamine-induced paroxysmal hypertension and normalize or reduce the exaggerated blood pressure variability in patients with familial dysautonomia (FD, also called hereditary sensory and autonomic neuropathy type III or Riley-Day syndrome). Funding Source- FDA OOPD.

DETAILED DESCRIPTION:
The investigators propose to perform a double-blind randomized trial with a cross over design to compare high dose (600 mg/day) and low dose (300 mg per day) carbidopa blockade with placebo. Patients will be randomly assigned to a high-dose/low-dose/placebo sequence, lowdose/placebo/high-dose sequence or placebo/high-dose/low-dose sequence. Participants will remain on each treatment period for 28-days.

Aim 1: To evaluate the safety and tolerability of carbidopa in FD patients with particular emphasis on the orthostatic fall in blood pressure.

Aim 2: As proof of concept, examine the hemodynamic effects of carbidopa and determine its effects on norepinephrine production, BP variability and paroxysmal hypertension.

Aim 3: In a dose finding study, compare the effects of low (300 mg/day) and high (600 mg/day) dose carbidopa blockade vs. placebo on BP variability and paroxysmal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with familial dysautonomia (FD) age 10 or older
* Unstable blood pressure, defined as:

  * Systolic BP standard deviation >15 mmHg
  * Or coefficient of variation >15%
  * Or documented episodic hypertensive peaks (>140mmHg)
* Confirmed diagnosis of FD (genetic testing)
* Providing written informed consent (or ascent) to participate in the trial
* Ability to comply with the requirements of the study procedures.

Exclusion Criteria:

* Patients taking monoamine oxidase (MAO)-inhibitors
* Patients taking: metoclopramide, domperidone, risperidone or other dopamine blockers
* Patients taking tricyclic antidepressants
* Patients taking neuroleptic drugs (haloperidol and chlorpromazine)
* Patients with a known hypersensitivity to any component of this drug.
* Patients with atrial fibrillation, angina or significant ECG abnormality
* Patients with significant pulmonary, cardiac, liver, renal (creatinine >2.0 mg/ml)
* Patients who have a significant abnormality on clinical examination that may, in the investigator's opinion might jeopardize their healthy participating in this trial.
* Women who are pregnant or lactating.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horacio C Kaufmann, MD, Principal Investigator — NYU School of Medicine; Lucy J Norcliffe-Kaufmann, PhD, Principal Investigator — NYU School of Medicine
Locations (2):
- United States (2):
  - NYU Langone Medical Center, Dyautonomia Center, Suite 9Q, New York, New York
  - NYU Medical Center, New York, New York

REFERENCES:
- [Background] Norcliffe-Kaufmann L, Martinez J, Axelrod F, Kaufmann H. Hyperdopaminergic crises in familial dysautonomia: a randomized trial of carbidopa. Neurology. 2013 Apr 23;80(17):1611-7. doi: 10.1212/WNL.0b013e31828f18f0. Epub 2013 Apr 3. PMID 23553478
- [Background] Norcliffe-Kaufmann LJ, Axelrod FB, Kaufmann H. Cyclic vomiting associated with excessive dopamine in Riley-day syndrome. J Clin Gastroenterol. 2013 Feb;47(2):136-8. doi: 10.1097/MCG.0b013e3182582cbf. PMID 22739220
- [Background] Norcliffe-Kaufmann L, Axelrod FB, Kaufmann H. Developmental abnormalities, blood pressure variability and renal disease in Riley Day syndrome. J Hum Hypertens. 2013 Jan;27(1):51-5. doi: 10.1038/jhh.2011.107. Epub 2011 Dec 1. PMID 22129610
- [Background] Kaufmann H, Malamut R, Norcliffe-Kaufmann L, Rosa K, Freeman R. The Orthostatic Hypotension Questionnaire (OHQ): validation of a novel symptom assessment scale. Clin Auton Res. 2012 Apr;22(2):79-90. doi: 10.1007/s10286-011-0146-2. Epub 2011 Nov 2. PMID 22045363
- [Background] Norcliffe-Kaufmann L, Axelrod F, Kaufmann H. Afferent baroreflex failure in familial dysautonomia. Neurology. 2010 Nov 23;75(21):1904-11. doi: 10.1212/WNL.0b013e3181feb283. PMID 21098405
- [Background] Palma JA, Norcliffe-Kaufmann L, Fuente-Mora C, Percival L, Mendoza-Santiesteban C, Kaufmann H. Current treatments in familial dysautonomia. Expert Opin Pharmacother. 2014 Dec;15(18):2653-71. doi: 10.1517/14656566.2014.970530. Epub 2014 Oct 17. PMID 25323828
- See also: New York University (NYU) Dysautonomia Center Research Site — http://med.nyu.edu/neurology/dysautonomia-center
- See also: Familial dysautonomia medical information — http://nyulangone.org/conditions/familial-dysautonomia
- See also: Patient Advocacy Group — http://familialdysautonomia.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-Dose Carbidopa, Then Placebo, Then High-Dose Carbidopa: Patients received low-dose carbidopa (300 mg/day), matching placebo, then high-dose carbidopa (600 mg/day) in 3 separate 4-week treatment periods. Doses were divided 3x daily, administered 6 hours apart, with a 4-day dose de-escalation and washout period between dose changes. in 3 separate 4-week treatment periods. Doses were divided 3x daily, administered 6 hours apart, with a 4-day dose de-escalation and washout period between dose changes.
- High-Dose Carbidopa, Then Low-Dose Carbidopa, Then Placebo: Patients received high-dose carbidopa (600 mg/day), low-dose carbidopa (300 mg/day), then matching placebo in 3 separate 4-week treatment periods. Doses were divided 3x daily, administered 6 hours apart, with a 4-day dose de-escalation and washout period between dose changes. in 3 separate 4-week treatment periods. Doses were divided 3x daily, administered 6 hours apart, with a 4-day dose de-escalation and washout period between dose changes.
- Placebo, Then High-Dose Carbidopa, Then Low-Dose Carbidopa: Patients received matching placebo, high-dose carbidopa (600 mg/day), then low-dose carbidopa (300 mg/day) in 3 separate 4-week treatment periods. Doses were divided 3x daily, administered 6 hours apart, with a 4-day dose de-escalation and washout period between dose changes.
Period: Enrollment
Arm/Group | Low-Dose Carbidopa, Then Placebo, Then High-Dose Carbidopa | High-Dose Carbidopa, Then Low-Dose Carbidopa, Then Placebo | Placebo, Then High-Dose Carbidopa, Then Low-Dose Carbidopa
Started | 9 | 7 | 6
Completed | 9 | 7 | 5
Not Completed | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Period: First Intervention (28 Days)
Arm/Group | Low-Dose Carbidopa, Then Placebo, Then High-Dose Carbidopa | High-Dose Carbidopa, Then Low-Dose Carbidopa, Then Placebo | Placebo, Then High-Dose Carbidopa, Then Low-Dose Carbidopa
Started | 9 | 7 | 5
Completed | 8 | 7 | 4
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Second Intervention (28 Days)
Arm/Group | Low-Dose Carbidopa, Then Placebo, Then High-Dose Carbidopa | High-Dose Carbidopa, Then Low-Dose Carbidopa, Then Placebo | Placebo, Then High-Dose Carbidopa, Then Low-Dose Carbidopa
Started | 8 | 7 | 4
Completed | 7 | 7 | 4
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Third Intervention (28 Days)
Arm/Group | Low-Dose Carbidopa, Then Placebo, Then High-Dose Carbidopa | High-Dose Carbidopa, Then Low-Dose Carbidopa, Then Placebo | Placebo, Then High-Dose Carbidopa, Then Low-Dose Carbidopa
Started | 7 | 7 | 4
Completed | 6 | 7 | 3
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Carbidopa, High Dose Carbidopa, Placebo: This is a 14-week study. Patients will receive, in random order, high dose carbidopa (600mg/day), low dose carbidopa (300 mg/day) or placebo. Between each crossover, there will be a titration down over 2-days followed by a 2-day washout.
  Carbidopa Low Dose
  Placebo: A placebo containing an inert substance, in capsule form that does not contain an active drug ingredient.
  Carbidopa High Dose
Arm/Group | Low Dose Carbidopa, High Dose Carbidopa, Placebo
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 28 [13 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Adverse Events Related to Study Drug
Description: Adverse events defined as: a change in a patient's baseline condition including intercurrent illnesses irrespective of the relationship to carbidopa treatment. This will be monitored primarily with phone calls at weekly intervals. In addition, patients will be asked about adverse events while at the office. Patients will also fill a daily diary with a specific prompts to note any adverse events.
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Low-Dose Carbidopa: 300 mg/day
  Other Names: Lodosyn ®, DL-α-methyl-α-hydrazino-3, 4-dihydroxyphenyl-propionic acid, HMD, MK-486
- High-Dose Carbidopa: 600 mg/day
  Other Names: Lodosyn ®, DL-α-methyl-α-hydrazino-3, 4-dihydroxyphenyl-propionic acid, HMD, MK-486
Arm/Group | Placebo | Low-Dose Carbidopa | High-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Significant Changes in Body Mass That Resulted in Discontinuation From the Study.
Description: Body mass measured in kg
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Low-Dose Carbidopa: 300 mg/day
  Other Name: Lodosyn ®, DL-α-methyl-α-hydrazino-3, 4-dihydroxyphenyl-propionic acid, HMD, MK-486
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Electrocardiographic Interval Patterns
Description: Clinically significant changes in the intervals of characteristic electrocardiographic patterns
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Groups:
- High-Dose Carbidopa: 600 mg/day
  Other Name: Lodosyn ®, DL-α-methyl-α-hydrazino-3, 4-dihydroxyphenyl-propionic acid, HMD, MK-486
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
Participants | 0 | 0 | 0

4. Primary Outcome: Average Systolic Blood Pressure Variability (Daytime)
Description: Patients with FD undergo ambulatory BP monitoring while keeping a detailed log of their activities (sleep/meal-times/medications/posture/symptoms). Variability in blood pressure overtime will be measured by the standard deviation during awake hours
Time Frame: up to Week 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
mmHg | 22.92 (6.13) | 18.71 (4.83) | 16.92 (4.14)

5. Primary Outcome: Highest Systolic Blood Pressure
Description: Maximum blood pressure captured on 24-h ambulatory monitoring
Time Frame: Day 1 of treatment period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
mmHg | 175 (27) | 157 (20) | 150 (17)

6. Primary Outcome: Systolic Blood Pressure
Description: SBP measured in the seated position
Time Frame: up to Week 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
mmHg | 126 (27) | 126 (18) | 126 (21)

7. Primary Outcome: Heart Rate
Description: Heart rate in the seated position
Time Frame: up to Week 14
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
beats per minute (BPM) | 76 (11) | 72 (13) | 78 (13)

8. Primary Outcome: Number of Participants Who Displayed Clinical Significant Laboratory Values on CBC or Metabolic Panel
Description: Clinically significant laboratory values include complete blood count (CMC) and metabolic panel related to treatment with carbidopa
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
Participants | 0 | 0 | 0

9. Primary Outcome: Number of Participants Who Displayed Clinically Significant Values in Urine Safety Parameters
Description: Clinically significant values on urinalysis, urine safety parameters related to treatment with carbidopa
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
Participants | 0 | 0 | 0

10. Secondary Outcome: Severity of Hypotension During an Active Stand Test
Description: Lowest blood pressure captured during 3 minutes of standing
Time Frame: up to Week 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
mmHg | 96 (27) | 91 (28) | 96 (24)

11. Secondary Outcome: Number of Participants Who Reported Worsening of OH Symptoms or Dropped Out Because of Worsening OH While on Active Study Drug
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
Participants | 0 | 0 | 0

12. Secondary Outcome: Frequency of Worsening Symptoms Noted in the Patient's Diary
Description: A tailored questionnaire to examine symptoms over the treatment period and the used of as needed medications. Each day will have a designated page. Since nausea/vomiting and hypertension occur together in FD we will use a diary consisting of a simplified version of the Rhodes Index 44 symptoms of nausea/retching, with items addressing vomiting/throwing up omitted, as most participants will have had anti-reflux surgery to prevent vomiting (fundoplication), graded on a 5-point scale (appendix 2). The diary will also include space to write down any adverse events on a daily basis.
Time Frame: Up to 90 Days
Measure: Number; unit: symptoms
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
symptoms | 0 | 0 | 0

13. Secondary Outcome: 24-h Urinary Norepinephrine Excretion
Description: Norepinephrine concentration determined from a 24-hour urine sample in a bottle shielded from light containing preservative. Patients will be instructed to refrigerate their sample and bring it on the morning of their visit in a cool bag.
Time Frame: up to Week 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
pg/mL | 16 (11) | 6 (3) | 8 (6)

14. Secondary Outcome: Coefficient of Systolic BP Variability (Daytime)
Description: The measurement of blood pressure variability based on the standard deviation that also takes into account the underlying level of BP.
Time Frame: up to Week 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
mmHg | 19 (4) | 16 (4) | 15 (3)

15. Secondary Outcome: Morning Surge in Systolic BP on Awakening From Sleep (24-h)
Description: The morning surge will be calculated as the difference between the mean systolic blood pressure during the hour that included the lowest blood pressure during sleep and maximum value detected within 2-h of awakening from sleep
Time Frame: up to Week 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | High-Dose Carbidopa | Low-Dose Carbidopa
Number analyzed (Participants) | 16 | 16 | 16
mmHg | 44 (24) | 19 (11) | 20 (9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Low-Dose Carbidopa | High-Dose Carbidopa | Placebo
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 3/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Carbidopa (N=16) | High-Dose Carbidopa (N=16) | Placebo (N=16)
Hospitaliztion (General disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-Dose Carbidopa (N=16) | High-Dose Carbidopa (N=16) | Placebo (N=16)
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 0
Syncope (Vascular disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT02553265/Prot_SAP_000.pdf